CLINICAL TRIAL: NCT04765254
Title: Clinical Features of Diabetic Patients With COVID-19 Infection
Brief Title: COVID-19 Infection in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia K. Zaafar, lecturer of pharmacology, Cairo University
Other Study IDs: ITH00131
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Diabete Type 2; Non Diabetic Patients; Chest CT Scan
Keywords: COVID-19; prognosis; mortality rate; Diabetes Mellitus
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samoles for routine CBC, D dimer and INR tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: COVID-19 infected patients with no other comorbidities and they take the routine protocol from the Egyptian ministry of health
  Interventions: Other: no intervention as it is an observational study
- diabetic group: COVID-19 infected patients with diabetes comorbidity and they receive the routine protocol for covid treatment in addition to their hypoglycemic drugs
  Interventions: Other: no intervention as it is an observational study

INTERVENTIONS:
Other: no intervention as it is an observational study — both groups will be monitored for the disease progress or deterioration and mortality rate

SUMMARY:
It was observed during the last period of COVID-19 pandemic that diabetic patients had a worse prognosis and more deteriorated clinical features than other patients

DETAILED DESCRIPTION:
Diabetic patients infected with SAR-COV-19 were reported to have worse prognosis and faster deterioration in addition to higher rate for ICU admission when compared to other infected patients. In this study authors aim to investigate the certain cause for their case deterioration to be modified for better prognosis

ELIGIBILITY:
Inclusion Criteria:

Patients infected with COVID-19 male or female 30 years old or more inpatients

Exclusion Criteria:

* have othe comorbidities other than type 2 diabetes mellitus pregnant women below 30 years old

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with COVID-19 either diabetic or have no comorbidities, inpatients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
Investigation of bad prognosis cause for covid-19 diabetic patients | 30 days
  number of diabetic patients with deteriorated case and to find the best hypoglycemic drug used for diabetic patients with covid-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University teaching hospitals, Cairo, Kasr Al Ainy, Egypt

IPD SHARING:
Plan to Share IPD: No